CLINICAL TRIAL: NCT00313703
Title: Predicting Poor Pain and Functional Outcomes After Discharge From the Emergency Department With a Primary Headache
Brief Title: Prospective ED Headache Cohort Study
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Prof. Emergency Medicine, Montefiore Medical Center
Other Study IDs: 04-03-077E
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Headache
Keywords: headache; emergency department; migraine; recurrent headache
MeSH Terms: conditions — Headache; Emergencies; Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine how often headaches recur and to learn how to predict continued suffering from headache after emergency department discharge.

DETAILED DESCRIPTION:
The majority of the 5 million people who arrive at Emergency Departments (ED) with a headache every year are suffering from an acute exacerbation of a chronic, recurrent headache disorder. The role of the ED in treating these patients has been ill-defined. Often emergency physicians will treat the acute exacerbation and will not attend to the natural history of the disease. However, about two thirds of primary headache patients will suffer a recurrent headache in the 24 hours after discharge from the ED. And, many patients will continue to suffer recurrent headaches for months after their ED discharge.

The purpose of this study is to learn how often headaches recur and to try to find a way to predict who will have a recurrent headache after ED discharge.

After standard ED treatment for headache, participants in the study will be asked to answer questions about prior headaches and medical history, and some census-like questions about race/ethnicity, salary, and education via a 20-minute interview with a research associate. The researchers will follow-up with 10-minute telephone calls to each participant's home in 24 hours and in 3 months with additional questions. Total length of time for study participation is approximately 40 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patients who present primarily for headache.
* Need to consent to and be available for follow-up

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience sample of ED patients
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2005-08 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, MS, Principal Investigator — Department of Emergency Medicine, Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, 111 East 210th Street, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled adult patients who presented to one urban emergency department (ED) with a chief complaint of headache.Patients were assigned a headache diagnosis based on criteria established by the International Headache Society (These are available at http://217.174.249.183/upload/CT_Clas/ICHD-IIR1final.pdf)
Pre-assignment Details: 477 patients underwent a detailed interview in the ED. 309 of these patients were determined to have a primary headache disorder (a benign recurrent headache disease) and were entered into the post-ED follow-up portion of this cohort study.
Groups:
- Migraine: met International Headache Society migraine criteria
- Tension-type Headache: met International Headache Society tension-type headache criteria
- Unclassifiable: Had recurrent headache disorder but did not meet any International Headache Society criteria
- Other: Met other International Headache Society criteria
Period: Overall Study
Arm/Group | Migraine | Tension-type Headache | Unclassifiable | Other
Started | 186 | 34 | 77 | 12
Completed | 175 (Some subjects lost to follow-up) | 32 (Some subjects lost-to follow-up) | 72 (Some subjects lost-to-follow-up) | 0 (Outcomes not reported due to heterogeneity of this group)
Not Completed | 11 | 2 | 5 | 12
Not completed — Lost to Follow-up | 11 | 2 | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Migraine | Tension-type Headache | Unclassifiable | Other | Total
Number analyzed (Participants) | 186 | 34 | 77 | 12 | 309
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38 (12) | 40 (12) | 42 (12) | 40 (11) | 39 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 25 | 54 | 8 | 256
  Male | 17 | 9 | 23 | 4 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Report Moderate or Severe Pain Within 24 Hours of Emergency Department(ED) Discharge
Description: Moderate/ Severe pain after discharge from the Emergency Department (ED). Moderate and severe are study subject's description of pain
Time Frame: 24 hours after Emergency Department (ED) discharge
Population: A small number of patients in each group were lost-to-follow-up and could not be included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Migraine | Tension-type Headache | Unclassifiable | Other
Number analyzed (Participants) | 172 | 32 | 75 | 0
Participants | 53 | 6 | 20 |

2. Other Pre Specified Outcome: Number of Participants Who Reported Headache Disability Scores (MIDAS) More Than Minimal
Description: Headache disability scores. On the MIDAS scale, a score > five signifies more than minimal headache related disability. MIDAS stands for MIgraine Disability Assessment Scale. More information on it can be found at http://www.migraines.org/disability/pdfs/midas.pdf. Scores of 0 are desirable. Scores greater than 20 signify a severe, functionally disabling migraine disorder.
Time Frame: 3 months
Population: A small number of patients in each group were lost-to-follow-up and could not be included in this analysis.
Measure: Number; unit: participants
Arm/Group | Migraine | Tension-type Headache | Unclassifiable | Other
Number analyzed (Participants) | 175 | 32 | 72 | 0
participants | 65 | 12 | 19 |

ADVERSE EVENTS:
Description: No adverse event information was gathered.
Arm/Group | Migraine | Tension-type Headache | Unclassifiable | Other
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No